CLINICAL TRIAL: NCT07177313
Title: Primary Ureteroscopy for Acute Obstructive Nephropathy Due to Ureteral Stones: A Prospective Non-randomized Feasibility and Safety Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mostafa Khedr, Residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Acute Obstructive Nephropathy
Record Dates: First submitted 2025-09-10; First posted 2025-09-16 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Acute Obstructive Nephropathy
MeSH Terms: interventions — Ureteroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Patients presenting with acute obstructive uropathy and uremic renal impairment (defined as serum creatinine ≥1.3 mg/dL)
  Interventions: Procedure: Ureteroscopy
- Group2 (Active Comparator): Patients with normal renal function (eGFR ≥60 mL/min/1.73m²) undergoing primary URS for ureteral stones.
  Interventions: Procedure: Ureteroscopy

INTERVENTIONS:
Procedure: Ureteroscopy — patients presenting with acute ureteral obstruction who undergo primary ureteroscopy (URS).

SUMMARY:
Ureteroscopy (URS) is a widely used minimally invasive procedure for the management of ureteral and renal stones (1). While the procedure is generally safe and effective, patient factors such as renal function, operative time, and ASA classification may influence outcomes (2).

Ureteral stones were found to be associated with deteriorated kidney function in affected patients (3). In cases of elevated urea and creatinine levels, pre-stenting of ureteroscopy was indicated (4). Limited number of studies have directly assessed the primary ureteroscopy without preoperative stenting outcomes in patients with normal versus deteriorated renal function. Understanding the impact of renal function on URS outcomes can help. A single procedure translates to reduced patient burden through fewer hospital visits, less time spent in the operating room, and a quicker return to daily activities, thus improving comfort and convenience. This approach also yields cost savings by eliminating the expenses associated with a second procedure, including hospital stays, anesthesia, and surgical supplies. Moreover, immediate stone removal via primary URS offers faster symptom relief and avoids potential stent-related complications such as pain, infection, and migration. However, the decision to forego staging must be carefully weighed against individual patient risk factors and stone complexity, as those with severe obstruction, infection, or compromised renal function may still benefit from pre-stenting to optimize procedural safety and outcomes.

This study aims to evaluate whether elevated creatinine levels influence stone-free rates, complication rates, and procedural success in patients undergoing primary URS.

ELIGIBILITY:
Inclusion Criteria:

* • Adults (>18 years) with acute unilateral ureteral obstruction confirmed by:
* Non-contrast CT (stone size ≥5mm)
* Hydronephrosis on ultrasound

  * Planned for primary URS (no prior stenting/nephrostomy)
  * Renal function eligibility:
* Acute deterioration (elevated serum Cr and urea) serum creatinine ≥1.3 mg/dL but less than 5 mg/dL

Exclusion Criteria:

• Systemic contraindications to URS:

* Uncorrected coagulopathy (INR >1.5)
* Active UTI/sepsis (requiring drainage-first approach)
* Severe cardiopulmonary compromise (ASA class ≥IV)

  * Patients with hypercalcemia.
  * hyperkalemia >6.5 mEq/L
  * Metabolic acidosis (pH <7.1)
  * Patients with pulmonary edema.
  * Patients with uremic encephalopathy.
  * Bilateral obstruction
  * Known ureteral stricture distal to stone

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
post operative complications | 3 month